CLINICAL TRIAL: NCT06570941
Title: A Pilot Study to Investigate the Benefits of a Cannabidiolic Acid Topical Cream for the Treatment of Restless Leg Syndrome
Brief Title: Benefits of a Cannabidiolic Acid Topical Cream for the Treatment of Restless Leg Syndrome
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Synthonics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHYLORLS-001
Record Dates: First submitted 2024-08-07; First posted 2024-08-26 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Intervention Model Description: therapeutic open label single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Benefits of a Cannabidiolic Acid Topical Cream for the Treatment of Restless Leg Syndrome (Experimental): Topical of application of cream to effected area 30-45 minutes before bedtime
  Interventions: Drug: Chylobinoid Topical Cream

INTERVENTIONS:
Drug: Chylobinoid Topical Cream — The topical cream is applied to the effected area to reduce or eliminate the symptoms of restless leg syndrome
  Other Names: Cannabidiolic acid topical cream

SUMMARY:
The goal of this open label clinical trial is to reduce the effects of restless leg syndrome. The main it questions it aims to answer are:

1. Reduce or eliminate the symptoms of restless leg syndrome.
2. Improve the quality of life of participants with restless leg syndrome.

Participants will be asked to apply the topical cream to the affected area 30 to 45 minutes before bedtime for 14 consecutive days.

DETAILED DESCRIPTION:
Restless Leg Syndrome (RLS) is multifactorial disease state with many different potential pathophysiological mechanisms, which includes dysfunctions from the cerebral cortex and spinal cord to mechanosensitive channels at the musculoskeletal periphery.1 Most therapeutic agents' effectiveness focuses on the CNS (e.g., dopaminergic drugs) or Renshaw cells. To our knowledge, therapeutic agents that are focused on the periphery were not very effective.

This technology focuses on the peripheral musculoskeletal component of the disease and is directed at treatment modalities that correct the dysfunction of mechanosensitive channels. By combining what is known about cannabinoids activity at the transient receptor potential channel of ankyrin 1 (TRPA1)2 and the role TRPA1 plays in regulating the shape and rigidity of the surrounding membrane structure at the Piezo channels3, an effective therapy at the site of discomfort should emerge. Moreover, the lessening of membrane tension is imparted by molecules that readily penetrate the membrane4, which Chylobinoid, the topical active ingredient, is uniquely designed to do.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 3 month-course of symptomatic restless leg syndrome
* Must meet International Restless Legs Syndrome Study Group (IRLSSG) criteria of at least mild symptoms.
* Age > 18 years, including both males and females
* Patient provides informed consent

Exclusion Criteria:

* Previous operative procedure for treatment of RLS;
* Current use of TENS (transcutaneous electrical nerve stimulation or plasma exchange;
* Allergy to Cannabidiol (CBD) Cannabidiolic acid (CBDa), or any other ingredient contained in the topical cream;
* Pregnant participants (participants who have the potential for being pregnant will sign a waiver), or breast feeding;
* History of recreational substance abuse, fibromyalgia, Chronic Regional Pain Syndrome (CRPS), psychiatric history including but not limited to schizoaffective disorder, bipolar disorder, chronic depression, and suicidal ideation;
* Conditions affecting capacity and adherence to study regimen including but not limited to dementia/delirium, Alzheimer's, Down's syndrome;
* A need for elective surgery involving preoperative or postoperative analgesics or anesthetics during the study period;
* No recent cannabinoid use in the last 2 months, and no use during the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Change of Restless Leg Syndrome | 14 days
  Severity of restless leg syndrome will be measured using the international restless leg syndrome questionnaire. It is a 10 question scale that is scored from 0 to 5 with 4 representing the most severe symptoms and 0 representing the least.

SECONDARY OUTCOMES:
Patient Quality of Life in response to treatment | 14 days
  Change measured by Patients' Global Impression of Change scale (PGIC). The scale is 3 to -2 with 3 being much improved and -2 being much worse.

CONTACTS AND LOCATIONS:
Locations (1):
- Synthonics, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romare, M., et al.
- [Background] De Petrocellis L, Vellani V, Schiano-Moriello A, Marini P, Magherini PC, Orlando P, Di Marzo V. Plant-derived cannabinoids modulate the activity of transient receptor potential channels of ankyrin type-1 and melastatin type-8. J Pharmacol Exp Ther. 2008 Jun;325(3):1007-15. doi: 10.1124/jpet.107.134809. Epub 2008 Mar 19. PMID 18354058
- [Background] Moparthi L, Zygmunt PM. Human TRPA1 is an inherently mechanosensitive bilayer-gated ion channel. Cell Calcium. 2020 Nov;91:102255. doi: 10.1016/j.ceca.2020.102255. Epub 2020 Jul 18. PMID 32717533
- [Background] Fang XZ, Zhou T, Xu JQ, Wang YX, Sun MM, He YJ, Pan SW, Xiong W, Peng ZK, Gao XH, Shang Y. Structure, kinetic properties and biological function of mechanosensitive Piezo channels. Cell Biosci. 2021 Jan 9;11(1):13. doi: 10.1186/s13578-020-00522-z. PMID 33422128
- [Background] Allen RP. Minimal clinically significant change for the International Restless Legs Syndrome Study Group rating scale in clinical trials is a score of 3. Sleep Med. 2013 Nov;14(11):1229. doi: 10.1016/j.sleep.2013.08.001. Epub 2013 Aug 14. No abstract available. PMID 24051118
- [Background] Piccariello, T., Palmer, S., Mulhare, M.; "Solid Micellar Compositions of Cannabinoid Acids"; International Application No. PCT/US2020/014109, filed January 17, 2020
- See also: Related Info — https://doi.org/10.5114/hm.2023.111547

DOCUMENTS (2):
  • Study Protocol (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT06570941/Prot_000.pdf
  • Informed Consent Form (2024-03-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT06570941/ICF_001.pdf